CLINICAL TRIAL: NCT07308990
Title: To Develop and Implement a Method for Optimizing the Volume of Lymph Node Dissection in Radical Surgical Treatment of Localized or Locally Advanced Prostate Cancer
Brief Title: Limited Versus Extended Lymph Node Dissection During Radical Prostatectomy in Patients With Localized or Locally Advanced Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Alexandrov National Cancer Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011/25
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy
Keywords: prostate cancer; lymph node dissection; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no / limited lymph node dissection (Experimental)
  Interventions: Procedure: Radical prostatectomy with limited / no lymph node dissection
- limited / extended lymph node dissection (Experimental)
  Interventions: Procedure: Radical prostatectomy with extended / limited lymph node dissection

INTERVENTIONS:
Procedure: Radical prostatectomy with extended / limited lymph node dissection — In patients with NCCN high or unfavorable intermediate risk prostate cancer - radical prostatectomy with extended lymph node dissection (incl. external iliac, obturator, internal iliac and common iliac nodes up to ureter bilaterally).
  In patients with NCCN low or favorable intermediate risk prostate cancer - radical prostatectomy with limited lymph node dissection (incl. obturator + / - external iliac lymph nodes bilaterally).
  Arms: limited / extended lymph node dissection
Procedure: Radical prostatectomy with limited / no lymph node dissection — In patients with NCCN high or unfavorable intermediate risk prostate cancer - radical prostatectomy with limited lymph node dissection (incl. obturator + / - external iliac lymph nodes bilaterally). In patients with NCCN low or favorable intermediate risk prostate cancer - radical prostatectomy with no lymph nodes dissection bilaterally.
  Arms: no / limited lymph node dissection

SUMMARY:
This is a randomized controlled study assessing outcome of low (no or limited) versus high (limited or extended) extent of lymph node dissection in addition to radical prostatectomy in patients with operable localized or locally advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Histologically confirmed localized or locally advanced prostate cancer (adenocarcinoma without a neuroendocrine component).
3. No evidence of metastatic spread of the tumor
4. Local resectability of the tumor according to digital rectal examination and/or CT and/or MRI of the pelvis
5. Patients are suitable for radical prostatectomy based on their comorbidities and life expectancy.
6. Signed informed consent to participate in the study.

Exclusion Criteria:

1. Presence of another active malignant invasive neoplasm.
2. Contraindication to pelvic lymph node dissection (e.g., history of radiation therapy to the pelvis).
3. The evidence of metastases in regional lymph nodes according to preoperative examination data (including PET/CT with PSMA).
4. Severe concomitant disease limiting participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2030-05-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | from enrollment to the end of the study at 5 years
  time from randomization to first diagnosis of distant metastasis from prostate cancer

SECONDARY OUTCOMES:
30-day complication rate | from the start of surgery to 30 days postoperatively
  rate of complications from the start of surgery to 30 days postoperatively graded by Clavien-Dindo
Perioperative events (length of surgery, intraoperative blood loss) | perioperatively
Duration of hospital stay | at first follow up visit (6-12 weeks post-surgery)
  time from surgery to the discharge from the hospital
Biochemical recurrence-free survival | from enrollment to the end of the study at 5 years
  time from randomization to first confirmed PSA rise > / = 0.2 ng/ml
Time to treatment | from enrollment to the end of the study at 5 years
  time from randomization to the first prostate cancer-related therapy
Prostate cancer specific survival | from enrollment to the end of the study at 5-7 years
  time from randomization to death from prostate cancer
Overall survival | from enrollment to the end of the study at 5-7 years
  time from randomization to to death of any cause
Metastasis-free survival in subgroups of patients (NCCN risk groups, operated by individual surgeon) | from enrollment to the end of the study at 5 years
  time from randomization to first diagnosis of distant metastasis from prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Alexandrov National Cancer Centre, Lyasny, Minsk Oblast, Belarus

IPD SHARING:
Plan to Share IPD: Undecided